CLINICAL TRIAL: NCT01624480
Title: A Randomized, Open-Label Study to Characterize the Pharmacokinetics, Pharmacodynamics, and Safety of Single and Multiple Doses of Armodafinil (50, 100, and 150 mg/Day) in Children and Adolescents With Excessive Sleepiness Associated With Narcolepsy
Brief Title: Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Safety of Armodafinil in Children and Adolescents With Excessive Sleepiness Associated With Narcolepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C10953/1100; 2012-005510-20 (EudraCT Number)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Narcolepsy
Keywords: Pediatric Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Armodafinil 50 mg (Experimental): In period 1, patients will receive a single 50-mg dose of armodafinil on day 1. In period 2, patients will receive a single 50-mg dose daily on days 1 through 42.
  Interventions: Drug: Armodafinil
- Armodafinil 100 mg (Experimental): In period 1, patients will receive a single 100 mg dose of armodafinil on day 1. In period 2, patients will receive a single 50-mg dose on day 1 then daily 100-mg doses on days 2 through 42.
  Interventions: Drug: Armodafinil
- Armodafinil 150 mg (Experimental): In period 1, patients will receive a single 150-mg dose of armodafinil on day 1. In period 2, patients will receive a single 50-mg dose on day 1, 100-mg doses on days 2 and 3, then daily 150-mg doses on days 4 through 42.
  Interventions: Drug: Armodafinil

INTERVENTIONS:
Drug: Armodafinil — The armodafinil tablets to be used in this study contain 50 mg of armodafinil and the following inactive ingredients: lactose monohydrate, starch, microcrystalline cellulose, croscarmellose sodium, magnesium stearate, and povidone.
  Other Names: R-modafinil; CEP-10953

SUMMARY:
This study is to evaluate the pharmacokinetics, pharmacodynamics, and safety of single and multiple doses of armodafinil (50, 100, and 150 mg/day) in children and adolescents with excessive sleepiness associated with narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained from each patient's parent or legal guardian and written assent is obtained from each patient.
* The patient is a male or female 6 through 17 years of age with a body mass index (BMI) equal to or greater than 10th percentile for age and gender, inclusive.
* The patient has a diagnosis of narcolepsy with cataplexy or narcolepsy without cataplexy according to the criteria established by the International Classification of Sleep Disorders (ICSD)-2 for narcolepsy.

Exclusion Criteria:

* The patient has any clinically significant uncontrolled medical condition (treated or untreated) other than narcolepsy.
* The patient has a clinically significant deviation from normal in ECG, physical examination or vital sign findings, as determined by the investigator or medical monitor.
* The patient is pregnant or lactating. (Any patient becoming pregnant during the study will be withdrawn from the study)
* The patient has any history of seizures, including febrile seizures, or a family history of seizures (in parents or siblings) which is not a consequence of trauma, stroke, or metabolic disturbance.
* The patient has a history of head trauma associated with loss of consciousness.
* The patient has current suicidal ideation, a history of a suicidal ideation, or a history of a suicide attempt.
* The patient has a history of major depressive disorder, bipolar disorder, other significant mood disorders, schizophrenia and other psychotic disorders, eating disorders, or has a family history of suicide.
* The patient has left ventricular hypertrophy or the patient has mitral valve prolapse and has experienced mitral valve prolapse syndrome.
* The patient has received any investigational drug within 30 days or 5 half-lives (whichever is longer) before the 1st dose of study drug, or in the case of a new chemical entity, 3 months or 5 half-lives (whichever is longer) before the 1st dose of study drug.

  * The patient has used any monoamine oxidase inhibitors (MAOIs) or stimulants within 14 days or 5 half-lives (whichever is longer) of the baseline visit.
  * The patient has used modafinil or armodafinil within 4 weeks of the baseline visit.
  * The patient has used an inducer of CYP3A4/5 within 28 days prior to study drug administration.
  * The patient has used an inhibitor of CYP3A4/5 within 14 days or 5 half lives (whichever is longer) prior to study drug administration.
  * The patient has a known sensitivity or idiosyncratic reaction to any compound present in modafinil or armodafinil, their related compounds, or to any metabolites or compound listed as being present in these medications.
  * The patient has a history of any clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reactions
  * Other criteria apply, please contact the investigator for additional information

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) by inspection | Day 1 + up to 72 hours after administration
Time to maximum observed plasma drug concentration (tmax) by inspection | Day 1 + up to 72 hours after administration
Area under the plasma drug concentration by time curve from time 0 to infinity | Day 1 + up to 72 hours after administration
Area under the plasma drug concentration by time curve from time 0 to the time of the last measurable drug concentration | Day 1 + up to 72 hours after administration
Terminal half-life | Day 1 + up to 72 hours after administration
Terminal elimination rate constant | Day 1 + up to 72 hours after administration
Apparent total plasma clearance | Day 1 + up to 72 hours after administration
Apparent volume of distribution | Day 1 + up to 72 hours after administration
Predicted accumulation ratio | Day 1 + up to 72 hours after administration
Maximum observed plasma drug concentration (Cmax) | Day 42 + up to 72 hours after administration
Time to maximum observed plasma drug concentration | Day 42 + up to 72 hours after administration
AUC over 1 dosing interval | Day 42 + up to 72 hours after administration
AUC 0-t | Day 42 + up to 72 hours after administration
Observed accumulation ratio | Day 42 + up to 72 hours after administration
Steady-state accumulation ratio | Day 42 + up to 72 hours after administration

SECONDARY OUTCOMES:
Mean sleep latency | 2 Days (Baseline + Day 1)
  An objective assessment of sleepiness that measures the likelihood of falling asleep. The test consists of multiple naps performed on the day before study drug administration in period 1 and on the day of study drug administration in period 1. For each nap, sleep latency will be measured as the elapsed time from lights-out to the first epoch scored as sleep. Mean sleep latency is calculated for each day as the average of the sleep latencies from each nap on that day.
Mean sleep latency | Day 42
  An assessment by the investigator of change in the patient's severity of excessive sleepiness during the course of the study. The clinician will ask the guardian to assess the child's home behavior over the past week.
Clinical Global Impression of Change (CGI-C) | Day 1
  An assessment by the investigator of change in the patient's severity of excessive sleepiness during the course of the study. The clinician will ask the guardian to assess the child's home behavior over the past week.
Clinical Global Impression of Change (CGI-C) | Outpatient Visits Weeks 1 through 5, once per week
  The Clinical Global Impression of Change (CGI-C) is an assessment by the investigator of change in the patient's severity of excessive sleepiness during the course of the study. The clinician will ask the guardian to assess the child's home behavior over the past week. The CGI-C ratings will be assessed using the following 7 categories and scoring assignments: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse
Clinical Global Impression of Change (CGI-C) | Day 42
  The Clinical Global Impression of Change (CGI-C) is an assessment by the investigator of change in the patient's severity of excessive sleepiness during the course of the study. The clinician will ask the guardian to assess the child's home behavior over the past week. The CGI-C ratings will be assessed using the following 7 categories and scoring assignments: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (24):
- United States (23):
  - Teva Investigational Site 12, Birmingham, Alabama
  - Teva Investigational Site 17, Birmingham, Alabama
  - Teva Investigational Site 7, Little Rock, Arkansas
  - Teva Investigational Site 18, Orange, California
  - Teva Investigational Site 16, San Diego, California
  - Teva Investigational Site 4, Stanford, California
  - Teva Investigational Site 9, Clearwater, Florida
  - Teva Investigational Site 26, Miami Lakes, Florida
  - Teva Investigational Site 5, Spring Hill, Florida
  - Teva Investigational Site 25, Winter Park, Florida
  - Teva Investigational Site 1, Atlanta, Georgia
  - Teva Investigational Site 2, Atlanta, Georgia
  - Teva Investigational Site 20, Louisville, Kentucky
  - Teva Investigational Site 15, Grand Blanc, Michigan
  - Teva Investigational Site 3, West Seneca, New York
  - Teva Investigational Site 23, Raleigh, North Carolina
  - Teva Investigational Site 10, Toledo, Ohio
  - Teva Investigational Site 13, Oklahoma City, Oklahoma
  - Teva Investigational Site 19, West Chester, Pennsylvania
  - Teva Investigational Site 8, Houston, Texas
  - Teva Investigational Site 14, San Antonio, Texas
  - Teva Investigational Site 27, Everett, Washington
  - Teva Investigational Site 24, Seattle, Washington
- Teva Investigational Site 200, Helsinki, Finland